CLINICAL TRIAL: NCT01828684
Title: Thin Film Spectacle Coatings to Reduce Light Sensitivity and Headaches in Patients With Migraine.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Katz (Other)
Responsible Party: Sponsor-Investigator, Bradley Katz, Associate Professor of Ophthalmology & Neurology, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB_00047263
Record Dates: First submitted 2013-04-07; First posted 2013-04-11 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Migraine Disorders; Photophobia
Keywords: Migraine with Aura; Migraine without Aura; Photophobia; Chronic Daily Headache
MeSH Terms: conditions — Migraine Disorders; Photophobia; Migraine with Aura; Migraine without Aura; Headache Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic Lens Coating (Experimental): Subjects will wear a therapeutic lens coating for 2 weeks
  Interventions: Other: Therapeutic Lens Coating; Other: Sham Lens Coating
- Sham Lens Coating (Sham Comparator): Subjects will wear a sham lens coating for 2 weeks
  Interventions: Other: Therapeutic Lens Coating; Other: Sham Lens Coating

INTERVENTIONS:
Other: Therapeutic Lens Coating — Subjects will wear a therapeutic lens coating for 2 weeks.
Other: Sham Lens Coating — Each subject will wear a sham lens coating for 2 weeks.

SUMMARY:
Approximately 9% of men and 18% of women suffer from migraine headaches. Almost all migraine sufferers report light sensitivity during a headache. Some people with migraine report that light can trigger their migraines and some people with migraine are light sensitive all of the time. The investigators have recently determined that certain colors of light are more likely to trigger migraines than other colors. In this study the investigators want to know if people who wear glasses that block these colors of light will have fewer migraine headaches.

ELIGIBILITY:
Inclusion Criteria:

1. Must be diagnosed with migraine with aura or migraine without aura
2. Must have chronic daily migraine (at least 15 headache days per month)
3. Age 18 or older

Exclusion Criteria:

1. Currently wearing a spectacle tint specifically prescribed for migraine or light sensitivity
2. Pregnant
3. Unwilling or unable in the judgment of the investigator to complete the study
4. Unavailable for any of the study visits
5. Light sensitive conditions: meningitis, iritis, blepharospasm
6. Degenerative diseases of the retina or optic nerve: diabetic retinopathy, ischemic optic neuropathy
7. Medications known to affect retinal or optic nerve function: hydroxychloroquine, chloroquine, ethambutol, amiodarone, erectile dysfunction drugs
8. Best corrected visual acuity less than 20/40 in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
HIT-6 | 10 weeks
  Primary outcome measure is improvement in HIT-6 while wearing therapeutic lenses compared to baseline. The HIT-6 is the Headache Impact Test, a trademarked and copyrighted test (2001 QualityMetric, Inc. and GlaxoSmithKline Group of Companies)

SECONDARY OUTCOMES:
Headache frequency and severity | 10 weeks
  Secondary outcome is reduction in headache frequency and severity as assessed by headache diaries.

OTHER OUTCOMES:
Photophobia | 10 weeks
  Tertiary outcome is reduction in photophobia as assessed by a photophobia questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J Katz, MD, Principal Investigator — University of Utah
Locations (1):
- John A Moran Eye Center; University of Utah Hospitals and Clinics, Salt Lake City, Utah, United States